CLINICAL TRIAL: NCT01065025
Title: Open Label, Dose Escalation Trial of Oral 4SC-205 in Patients With Advanced Malignancies: First-In-Man Study of a Newly Developed, Oral Inhibitor of Kinesin-spindle Protein, Eg5
Brief Title: Open Label, Dose Escalation Trial of Oral Eg5 Kinesin-spindle Inhibitor 4SC-205 in Patients With Advanced Malignancies
Acronym: AEGIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4SC AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-205-1-2009
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Advanced and Incurable Solid Tumors; Malignant Lymphomas
Keywords: 4SC-205; Solid tumors; Lymphomas; Phase I
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 4SC-205 (Experimental)
  Interventions: Drug: 4SC-205

INTERVENTIONS:
Drug: 4SC-205 — Repeated ascending oral doses of 4SC-205.

SUMMARY:
The purpose of the study is to investigate safety and tolerability of repeated ascending oral doses of 4SC-205 in patients with advanced and incurable solid tumors or malignant lymphomas.

ELIGIBILITY:
Main Inclusion Criteria:

* One or more evaluable target lesion according to RECIST (by CT-scan, MRI or calipers), of which at least one evaluable target lesion (proven by CT or MRI) has to be located in the lung.
* Progressive disease as defined by new or progressive lesions on CT-scan, MRI, bone scan or by increase of PSA.
* Histologically or cytologically documented diagnosis of primary or metastatic solid tumors or malignant lymphomas refractory to prior standard therapy or for which no standard therapy exists. Entry will include, but is not limited to patients with prostate and breast cancer refractory to hormone treatment, ovarian cancer, head and neck cancer, non-small cell lung cancer, bladder cancer, colorectal cancer, kidney cancer, malignant melanoma or malignant lymphoma. Patients who have refused standard therapies are also eligible.
* ECOG Performance Status 0-2.
* Acceptable liver, renal and bone marrow function.

Main Exclusion Criteria:

* Prior treatment with other EG5 inhibitors.
* Antineoplastic therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the last 2 weeks or a longer period depending on the defined characteristics of the agents used (e.g. 6 weeks for mitomycin C or nitrosourea). Patients must have recovered from any treatment-related toxicity (except for alopecia, fatigue and grade 1 neurotoxicity) prior to registration.
* Patients with a history of other malignancies unless having undergone definitive treatment more than 5 years prior to entry into the study and without evidence of recurrent malignant disease, excluding patients with basal cell carcinoma of the skin; superficial carcinoma of the bladder; carcinoma of the prostate with a current PSA < 0.1 ng/ml; or cervical intraepithelial neoplasia.
* Patients with a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory or inflammatory illness.
* Patients with a history of, who were treated for, or who are suspected of having, hepatitis B, hepatitis C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of repeated ascending oral doses of 4SC-205. Determination of the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT). | 6 weeks

SECONDARY OUTCOMES:
Pharmacokinetics | 6 weeks
Anti-cancer activity of 4SC-205 after 6 weeks of treatment. | 6 weeks
Effects of EG5 inhibition on biomarker modulation. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mross, PD Dr. med., Principal Investigator — Klinik für Tumorbiologie an der Albert-Ludwigs-Universität Freiburg (KTB)
Locations (2):
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Klinik für Tumorbiologie an der Albert-Ludwigs-Universität Freiburg (KTB), Freiburg im Breisgau